CLINICAL TRIAL: NCT07233174
Title: Postprandial Thermogenesis in Obese Adolescents: Effect of Meal Calorie Content
Acronym: TEFAO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Emile Roux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RIPH2_GADEA_TEFAO; 2025-A01847-42 (Other: ID RCB)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Obesity (Disorder)
Keywords: obesity
MeSH Terms: conditions — Obesity | interventions — Energy Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescents aged 11 to 17 with obesity (Experimental)
  Interventions: Other: Energy expenditure and energy substrates; Other: Food sensations; Other: Liking & Wanting

INTERVENTIONS:
Other: Energy expenditure and energy substrates — * Three randomized experimental visits to the AME2P laboratory with a minimum interval of five days between each visit with:
  * one test meal with a different calorie content but the same macronutrient distribution: i) a 700 kcal meal (C-700); ii) a 1000 kcal meal (C-1000); iii) a 1300 kcal meal (C-1300).
  * Energy expenditure and energy substrates: at the adolescents' arrival at the laboratory (20 min), then for 20 min before the test meal at noon, then for one hour immediately after the meal, then for 15 min every 45 min after the meal for 4 hours.
  Mesured using portable indirect calorimetry (MetaMax, Inc.).
Other: Food sensations — At regular intervals throughout the experimental days, participants will be asked to complete visual analog scales (VAS) to report their feelings of hunger, satiety, or desire to eat. Measurements will be taken before and after breakfast, same for the test lunch, and then every 30 min until 5 p.m.
Other: Liking & Wanting — Their relationship with food will be investigated 15 min before the test meal and then 1 hour after, using the Leeds Foods Preference Questionnaire developed and validated by the team led by Professor Blundell. The adolescents will be asked to answer a series of questions about their food preferences by selecting their favorite foods from a selection of images during a 10-min computer exercise. Similarly, during this exercise, they are asked to use a visual analog scale to estimate how much they would like to eat certain foods presented. Based on their choices and the time taken to respond, the LFPQ assesses the adolescents' degree of "liking" and "wanting." The adolescents must complete this exercise 15 minutes before and after the evening test meal. To avoid any influence on food intake at the next meal, the foods presented during the test are not foods presented during the meal. The objective of this exercise is to assess the response of "liking" and "wanting" to food intake.

SUMMARY:
The prevention and management of pediatric obesity require a thorough understanding and consideration of the different components of energy balance (i.e., intake and expenditure) and their interactions. Total energy expenditure (TEE) consists of resting metabolism (RM), energy expenditure induced by physical activity (EEPA), and dietary thermogenesis (DTE). While RM and EEPA are the two main contributors to TEE, DTE is often overlooked, even though it can account for around 10% of our daily energy expenditure. In fact, few studies have prioritized the evaluation of the thermic effect of food (TEF), defined as the increase in energy expenditure above the basal metabolic rate when fasting, despite the fact that it accounts for about 10% of total daily energy expenditure . It has been suggested that TEF may play a role in the development or maintenance of obesity.

Some studies indicate a reduction in TEF in individuals living with obesity , possibly due to lower postprandial activation of the sympathetic nervous system, thereby limiting the thermogenic response after meals . Conversely, several studies have reported no decrease in TEF in individuals living with obesity . Due to these contradictory results, no consensus has been reached on the FET response in individuals with obesity compared to those of normal weight.

The limited number of available results can be explained not only by a lack of interest in this TEF among scientists and clinicians, but also by the methodological difficulties involved in its assessment. Indeed, the latter requires indirect calorimetry measurements over a period of up to 5 to 6 hours after a meal, as well as careful calibration of the test meals used, their qualitative content, and their caloric content. These factors are all the more important to consider given that a systematic review has shown that TEF is influenced by the energy intake of the meal as well as its macronutrient composition, with proteins and carbohydrates inducing a higher TEF than lipids . However, several uncertainties remain, particularly regarding the choice of test meal, which could be standardized for all participants or adjusted according to their body composition.

While our team recently conducted a systematic review of the literature in this area, identifying a glaring lack of evidence, the few results available suggest a potential reduction in TEF in obese children and adolescents, contributing to a minimization of the optimization of their daily energy balance. In their study, Maffeis and colleagues show, for example, a significantly reduced TEF in adolescents with obesity compared to their normal-weight counterparts, despite a higher-calorie test meal adapted to their energy needs . These results are consistent with those proposed by Salas-Salvado the following year, who suggested a reduced TEF in obese adolescents, associated with their percentage of body fat . This research suggests the need to consider the effects of weight status, body composition, and the caloric composition of a meal in order to better understand TEF in this population.

Unfortunately, this area has not been explored in depth since the 1990s, even though the prevalence of pediatric obesity continues to rise.

In this context, the objective of this study is to explore dietary thermogenesis in response to meals of different caloric content in obese adolescents.

ELIGIBILITY:
Inclusion Criteria:

* • Adolescents aged 11 to 17 (inclusive), at Tanner stage 3-5 of sexual maturation,

  * With obesity defined as a body mass index (BMI) above the 97th percentile according to national growth charts,
  * Adolescents affiliated with the social security system or equivalent,
  * Adolescents who have been informed and have given their written consent to participate in the study.

Exclusion Criteria:

* Refusal to participate in the study,
* Refusal of consent by legal guardians,
* Regular consumption of tobacco or alcohol,
* Special diet,
* Participation in regular and intense physical and sporting activities,
* Medical or surgical history deemed by the investigator to be incompatible with the study,
* Presence of diabetes, and any other condition limiting the application of either strategy being tested,
* Adolescents undergoing energy restriction or a weight loss program through physical activity at the time of inclusion or during the last 6 months,
* Taking medication that may interfere with the study results.
* Adolescents with cardiovascular problems, i.e., subjects with a history of cardiovascular and/or neurovascular disease, as well as subjects with cardiovascular and/or neurovascular risk factors (excluding obesity/overweight).
* Surgery in the previous 3 months,
* Adolescents who are currently excluded from another study,
* Pregnant or breastfeeding adolescents,
* Adolescents under guardianship/curatorship or legal protection,
* Parents under guardianship/curatorship or legal protection.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2025-12-03 (Actual); Primary Completion 2026-01-21 (Actual); Study Completion 2026-01-21 (Actual)

PRIMARY OUTCOMES:
Postprandial energy expenditure (PEE) in response to meals. | Visit 1, Visit 2, Visit 3
  Energy expenditure and energy substrates will be assessed in the morning upon arrival at the laboratory (20 minutes), then for 20 minutes before the test meal at noon, then for one hour immediately after the meal, then for 15 minutes every 45 minutes after the meal for 4 hours (a total of 5 hours of post-meal measurements).
  These measurements will be performed using portable indirect calorimetry (MetaMax, Inc.). Indirect calorimetry is one of the classic methods for measuring resting energy expenditure . The contribution of lipid and carbohydrate oxidation will be calculated indirectly by monitoring oxygen consumption and CO2 rejection according to double unknown equations, considering that protein oxidation is stable and around 15% .
  The MetaMax is a mask that causes no physical or respiratory discomfort and is connected to a gas analyzer. This technology has been used regularly in adolescents with and without obesity by our team and other teams .

SECONDARY OUTCOMES:
Appetite sensations in response to meals | Visit 1, Visit 2, Visit 3
  At regular intervals throughout the experimental days, participants will be asked to complete Visual Analog Scales to report their feelings of hunger, satiety, or desire to eat. Measurements will be taken before and after breakfast, before and after the test lunch, and then every 30 minutes until 5 p.m.
  Participants will be asked questions such as, if hungry or not, and will quantify their feelings on a scale of 0mm to 150mm, with 0mm corresponding to the minimum and "Not at all" and 150mm to the maximum and "Extremely." These scales, proposed and validated by Flint and colleagues in 2001 (Flint Scale), have been used in adults and children, both thin and obese, and have shown high reliability of results.
The hedonic response as measured by food liking and wanting | Visit 1, Visit 2, Visit 3
  The study examines adolescents' relationship with food using the Leeds Food Preference Questionnaire. During a 10-minute computer task, participants choose preferred foods from images and rate how much they would like to eat each item using visual analogue scales. Their reaction times and ratings allow researchers to measure both "liking" and "wanting." The task is completed 15 minutes before and after the evening test meal, and the foods shown differ from those served to avoid influencing intake. Liking is rated on a scale from 0 ("not pleasant at all") to 100 ("extremely pleasant"), with higher scores indicating stronger liking. Wanting is measured on a similar scale from 0 ("do not want at all") to 100 ("strongly want to eat"), where higher scores reflect greater motivational desire for the food.

CONTACTS AND LOCATIONS:
Overall Officials: David THIVEL, Principal Investigator — Director of AME2P Laboratory, Clermont Ferrand
Locations (1):
- Laboratory AME2P, University of Clermont Auvergne, Aubière, France